CLINICAL TRIAL: NCT07388004
Title: Rewiring Expectations and Amplifying Rewards: A Study Protocol for a Randomized Controlled Trial of Mechanism-Based Group Psychotherapy for Major Depressive Disorder
Brief Title: Group Therapy for Major Depression: Comparing Expectation-Focused and Reward-Focused Psychotherapy Approaches
Acronym: PERSPECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERSPECT CRC393-C02; 521379614 (Other Grant/Funding Number: German Research Foundation (Deutsche Forschungsgemeinschaft, DFG)); 23-272BO (Other: Ethics Committee of Philipps-University Marburg)
Record Dates: First submitted 2025-12-08; First posted 2026-02-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; Psychotherapy; Group Therapy; Expectation Violation; Reward Sensitivity; Mechanism-Based Intervention; Randomized Clinical Trial
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in equal proportions to one of three parallel groups: EFPI, REACT, or waiting-list control.
Who Masked: Outcomes Assessor
Masking Description: Independent outcome assessors conducting clinician-rated measures (e.g., HAMD-21) will remain blinded to group allocation. Participants, therapists, and investigators are not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Expectation-Focused Psychotherapeutic Intervention (EFPI) (Experimental): Participants receive 10 group therapy sessions (2 sessions per week over 5 weeks) of EFPI, a mechanism-based psychotherapy targeting maladaptive expectations.
  The intervention combines psychoeducation, structured behavioral experiments, and cognitive restructuring to systematically challenge negative expectations.
  A central focus is reducing cognitive immunization-the tendency to dismiss or reframe positive disconfirming evidence-to foster more flexible and adaptive belief updating.
  Sessions are conducted in small groups (5-10 participants) to facilitate peer modeling, social reinforcement, and shared learning.
  The first session includes baseline clinical assessments, and the final session includes immediate post-treatment assessments.
  All participants are additionally followed up at 3 and 6 months after the intervention to evaluate the persistence of treatment effects.
  Interventions: Behavioral: Expectation-Focused Psychotherapeutic Intervention
- Reward Enhancement and Activation Therapy (REACT) (Experimental): Participants receive 10 group therapy sessions (2 sessions per week over 5 weeks) of REACT, a mechanism-based psychotherapy designed to enhance reward sensitivity.
  Core intervention components include attentional retraining toward rewarding stimuli, savoring exercises to prolong positive affect, and structured reinforcement plans to strengthen motivation and engagement in rewarding activities.
  Group discussions normalize difficulties in experiencing pleasure and provide strategies for sustaining rewarding behavior long-term.
  Sessions are conducted in small groups (5-10 participants). The first session includes baseline assessments, and the final session includes immediate post-treatment assessments.
  Long-term outcomes are assessed through follow-up evaluations at 3- and 6-months post-intervention.
  Interventions: Behavioral: Reward Enhancement and Activation Therapy
- Waiting-List Control (No Intervention): Participants assigned to the waiting-list control condition do not receive active treatment during the initial 3-month period.
  They complete baseline assessments at study entry and a follow-up assessment after 3 months, corresponding to the time frame of the active intervention arms.
  After the 3-month assessment, participants are ethically permitted to pursue standard care outside the study.
  For comparability and long-term analyses, waiting-list participants continue to complete follow-up assessments at 6 months, including questions about any additional treatments received after the waiting-list phase.

INTERVENTIONS:
Behavioral: Expectation-Focused Psychotherapeutic Intervention — EFPI is a manualized group psychotherapy for major depressive disorder that directly targets maladaptive expectations. The treatment integrates psychoeducation, cognitive restructuring, and behavioral experiments to modify negative expectancies and reduce cognitive immunization, thereby enhancing adaptive expectation updating.
  Delivery: Group format (5-10 participants), 10 sessions (twice weekly for 5 weeks).
  Other Names: EFPI
  Arms: Expectation-Focused Psychotherapeutic Intervention (EFPI)
Behavioral: Reward Enhancement and Activation Therapy — REACT is a manualized group psychotherapy for major depressive disorder that focuses on enhancing reward sensitivity and motivation. The intervention combines attentional retraining, savoring techniques, and reinforcement-based strategies to increase engagement with rewarding stimuli and experiences.
  Delivery: Group format (5-10 participants), 10 sessions (twice weekly for 5 weeks).
  Other Names: REACT
  Arms: Reward Enhancement and Activation Therapy (REACT)

SUMMARY:
Major depressive disorder (MDD) is one of the most common psychiatric conditions and often remains difficult to treat effectively. Many patients continue to experience residual symptoms or relapse even after receiving established forms of psychotherapy. This study tests whether targeting specific psychological mechanisms can improve outcomes for people with depression. We compare two novel group therapies: (1) Expectation-Focused Psychotherapeutic Intervention (EFPI), which aims to modify rigid, negative expectations that maintain depressive symptoms, and (2) Reward Enhancement and Activation Therapy (REACT), which focuses on increasing sensitivity to positive experiences and strengthening reward-related learning. Both are delivered in a group format to foster peer support and shared learning.

A total of 150 adults with a current MDD diagnosis will be randomly assigned to EFPI, REACT, or a waiting-list control. Participants in the intervention groups receive 10 group sessions over five weeks. Waiting-list participants complete baseline and 3-month follow-up assessments before being offered standard treatment options.

Clinical outcomes are assessed at baseline, immediately after treatment, and at 3- and 6-month follow-ups (for the intervention groups). Primary outcomes are reductions in depressive symptoms measured by clinician ratings and self-report questionnaires. Secondary outcomes include changes in expectation processes and reward sensitivity.

In addition, functional MRI (fMRI) tasks examine brain mechanisms related to expectation updating and reward processing pre- and post-intervention, to help identify neural changes that may underlie symptom improvement.

By directly addressing dysfunctional expectations and reduced reward sensitivity, this study seeks to provide evidence for more targeted psychotherapeutic approaches. If successful, the results may support more personalized treatments and better long-term outcomes in MDD.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) remains a leading cause of disability and often shows incomplete response or relapse after established treatments. A promising strategy is to move beyond broad, symptom-focused interventions toward therapies that directly target the psychological and neurobiological mechanisms maintaining depression. This trial evaluates two mechanism-based, group-delivered psychotherapies that each target a core process implicated in MDD: maladaptive expectation processing and reduced reward sensitivity.

Rationale and mechanistic framework. Expectation pathway. Predictive coding accounts propose that the brain continuously updates prior beliefs in light of new information. In depression, negative expectations about the self, others, and the future often become rigid and resistant to change. Cognitive immunization-discounting or reframing disconfirming evidence-prevents adaptive belief updating, maintains symptoms, and can weaken responses to conventional cognitive-behavioral interventions. Targeting dysfunctional expectations directly-via structured behavioral experiments that produce positive expectation violations and procedures that reduce cognitive immunization-may restore flexibility in belief revision and enhance treatment effects.

Reward pathway. Depressed patients frequently show reduced reward sensitivity, including blunted anticipation of reward and impaired reinforcement learning, processes linked to mesolimbic dopaminergic circuitry (e.g., ventral striatum/nucleus accumbens). These deficits can limit the benefit of nonspecific activity scheduling, which increases exposure to potentially rewarding situations but does not specifically remediate anticipatory and learning-related components of reward processing. Interventions that systematically enhance reward sensitivity and strengthen reinforcement contingencies may therefore improve motivational drive and positive affect.

Neurobiological component. Expectation updating has been associated with activity in the dorsolateral prefrontal cortex (DLPFC) and anterior insula, whereas reward processing consistently engages the ventral striatum and insular cortex. This trial includes a functional MRI (fMRI) module to probe these mechanisms pre- and post-intervention. Participants perform established paradigms tapping threat/expectation learning, future-directed thinking, and social reward/expectation. Linking neural responses to clinical change will clarify how mechanism-based therapies exert their effects and may inform biomarkers for treatment selection and monitoring.

Study design overview. This is a randomized, controlled, superiority trial with three parallel groups: (1) EFPI, (2) REACT, and (3) waiting-list control. The trial follows a 3 × 5 repeated-measures design with planned assessments at baseline (pre-treatment), post-treatment (after 5 weeks), and 3- and 6-month follow-ups. Intervention groups complete all follow-ups; after the 6-month assessment they may initiate further treatment if desired. Waiting-list participants complete baseline and the 3-month follow-up before being ethically permitted to access other treatments. They continue to receive follow-up questionnaires at later time points, including items on additional treatments, to enable sensitivity analyses.

Randomization is performed at the individual level with a 1:1:1 allocation ratio. Allocation is managed through secure electronic data capture to ensure concealment until assignment. Given the nature of group psychotherapy, participants and therapists are not blinded; however, outcome assessors remain blind to group allocation, and standardized procedures are applied for clinician-rated measures. Because treatment is delivered in groups, potential therapist- and group-related effects are monitored and considered analytically.

Interventions (concise). EFPI and REACT are manualized group interventions delivered in 10 sessions over five weeks (two 100-minute sessions per week) by trained CBT therapists under regular supervision.

* EFPI targets maladaptive expectations and cognitive immunization through psychoeducation; identification/documentation of negative expectations; structured real-life behavioral experiments (predict-test-experience-reflect); guided cognitive integration to promote flexible belief updating; and maintenance strategies.
* REACT targets reduced reward sensitivity through systematic reinforcement procedures: identifying reward deficits and attentional biases; enhancing and prolonging positive experiences (e.g., savoring, imagery); structured engagement in meaningful rewarding activities with explicit reinforcement plans; and relapse-prevention strategies to sustain reward engagement.

Therapist training, supervision, adherence checklists, and standardized materials support fidelity. The waiting-list control receives no active group intervention during the first three months but is offered standard treatment options thereafter.

Assessments and timeline (overview). Clinical and behavioral data are collected at baseline, post-treatment, 3- and 6-month follow-ups in the intervention arms; the waiting-list control is assessed at baseline and 3 months prior to accessing further care. Digital data capture (e.g., REDCap) includes automated range and plausibility checks; follow-ups are facilitated via secure online questionnaires and structured telephone contacts to minimize attrition. In addition to clinician- and self-rated depression severity, the battery includes validated measures of expectation processing, reward sensitivity (anticipatory and learning components), and related cognitive-emotional constructs. Eligibility criteria and outcome measures are specified elsewhere in this record.

Neuroimaging component (overview). An fMRI module is acquired at baseline and post-intervention (or the matched 3-month time point for the waiting-list group) to assay neural correlates of expectation updating and reward processing. Paradigms include: (i) conditioning-based tasks probing threat expectancy and expectation violation; (ii) future-directed thinking tasks eliciting positive/negative prospective/retrospective imagery; and (iii) a social reward/expectation paradigm using structured interactions with virtual partners. Region-of-interest analyses focus on DLPFC/anterior insula (expectation) and ventral striatum/insula (reward); whole-brain and connectivity analyses complement ROI findings. Standard preprocessing (e.g., motion correction, normalization, smoothing) and task-based GLMs with multiple-comparison control are used. Neuroimaging endpoints are related to clinical trajectories to test mechanistic hypotheses.

Adherence, concomitant care, and retention. Participants confirm availability for the 5-week schedule before enrollment; attendance is monitored and automated reminders are sent. During the 5-week intervention phase, participants are asked to maintain stable psychotropic medication and to refrain from initiating additional psychotherapy; deviations are documented. After the intervention, participants may seek external psychotherapy; additional treatments at follow-up are recorded for sensitivity/covariate analyses. Retention is supported through reminders, flexible scheduling, and brief telephone assessments if full questionnaires are declined.

Sample size and operating characteristics. Planned enrollment is N = 150 (~50 per arm), allowing for expected attrition while preserving power to detect group × time effects of practical relevance in linear mixed-effects models. Power considerations were based on moderate effects from prior mechanism-focused psychotherapy literature; primary analyses will use linear mixed models.

Statistical analysis (overview). Primary clinical analyses use linear mixed-effects models with fixed effects for Group, Time, and their interaction, and random intercepts (and where appropriate, random slopes) to account for within-subject dependency and between-subject heterogeneity. Models will consider therapist/group clustering where indicated. Prespecified mediation analyses test whether changes in expectation processing and reward sensitivity account for symptom change; moderation analyses examine whether baseline profiles predict differential benefit. Missing data are handled under missing-at-random assumptions using maximum likelihood, with multiple imputation in sensitivity analyses. Neuroimaging analyses relate pre-to-post changes in activation/connectivity to clinical improvements; ROI-based hypotheses are complemented by exploratory whole-brain analyses with appropriate error control.

Safety monitoring and harms. Given the non-invasive, low-risk nature of group psychotherapy, no independent Data Safety Monitoring Board is planned. Safety is monitored by the investigative team throughout treatment and follow-up. Adverse events (including clinically significant symptom worsening or emergent suicidality) are documented and managed according to predefined procedures, with referral to appropriate care as needed and ethics notification when required. Criteria for discontinuation include persistent non-attendance or need for higher-level care during the intervention phase.

Data management and confidentiality. All data are pseudonymized (unique study IDs); identifying information is stored separately on access-restricted institutional servers. Electronic data capture uses role-based access, audit trails, and automated checks. After completion, personally identifying data are deleted; anonymized datasets are retained per policy and may be shared under GDPR-compliant agreements to support transparency and reproducibility.

Ethical conduct and dissemination. The protocol adheres to SPIRIT recommendations and has received ethics approval from the responsible institutional review board. Written informed consent is obtained from all participants prior to any study procedures. Results will be disseminated via peer-reviewed publications and scientific meetings; de-identified data and analysis code may be shared under controlled access agreements to promote open science.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years
* Current diagnosis of major depressive disorder (MDD) according to DSM-5, confirmed by structured clinical interview (e.g., DIPS)
* Hamilton Depression Rating Scale (HAMD-21) score ≥ 9
* Ability to attend group therapy sessions (2×/week for 5 weeks)
* Ability to undergo MRI scanning (for participants in the fMRI component) Written informed consent

Exclusion Criteria:

* Current or lifetime diagnosis of bipolar disorder, psychotic disorder, or primary substance use disorder
* High acute suicide risk requiring immediate intervention
* Severe neurological disorder, brain injury, or contraindications for MRI (e.g., metal implants, claustrophobia)
* Ongoing psychotherapy or initiation of a new antidepressant medication within the past 4 weeks
* Insufficient German language proficiency to participate in therapy and complete study assessments
* Cognitive impairment or other conditions interfering with informed consent or study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms (Beck Depression Inventory-II) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in depressive symptom severity assessed with the Beck Depression Inventory-II (BDI-II), a 21-item self-report questionnaire measuring cognitive, affective, and somatic symptoms of depression.
  Total scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
  The primary endpoint is the change from baseline to post-treatment (5 weeks). Symptom stability and maintenance will be examined at follow-up assessments.

SECONDARY OUTCOMES:
Change in Depressive Symptoms (Hamilton Depression Rating Scale, 21-item) | Baseline and post-treatment (5 weeks)
  Change in clinician-rated depressive symptom severity assessed with the Hamilton Depression Rating Scale (HAMD-21), administered by trained, blinded assessors.
  Total scores range from 0 to 64, with higher scores indicating more severe depressive symptoms.
Depressive Expectations (Depressive Expectations Scale) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in depressive expectations assessed with the Depressive Expectations Scale (DES), a self-report questionnaire measuring negative, situation-specific expectations related to mood regulation, social interactions, performance, and coping. Items are rated on a 5-point Likert scale; higher scores indicate more negative and dysfunctional expectations.
Hopelessness (Beck Hopelessness Scale) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in hopelessness assessed with the Beck Hopelessness Scale (BHS), a 20-item self-report questionnaire measuring negative expectations about the future.
  Total scores range from 0 to 20, with higher scores indicating greater hopelessness.
Socially Negative Expectations (Social Anxiety-Negative Beliefs Scale, SANB-5) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in negative social expectations assessed with the Social Anxiety-Negative Beliefs Scale (SANB-5), a 5-item self-report measure capturing fears of negative evaluation and rejection in social contexts.
  Items are rated on a 4-point Likert scale; higher scores indicate stronger negative social expectations.
Behavioral Activation and Reward Responsiveness (Behavioral Activation System Scale) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in reward responsiveness assessed with the Behavioral Activation System (BAS) Scale, a self-report questionnaire measuring approach motivation, reward sensitivity, and positive affective reactivity.
  Items are rated on a 4-point Likert scale; higher scores indicate greater behavioral activation and reward sensitivity.
Resilience (Resilience Scale, RS-25) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in psychological resilience assessed with the Resilience Scale (RS-25), a 25-item self-report questionnaire measuring personal competence, acceptance of self and life, and adaptive functioning.
  Items are rated on a 7-point Likert scale; higher scores indicate greater resilience.
General Self-Efficacy (Allgemeine Selbstwirksamkeit Kurzskala, ASKU) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Change in perceived self-efficacy assessed with the General Self-Efficacy Short Scale (ASKU), a 3-item self-report measure of confidence in one's ability to cope with difficult situations.
  Items are rated on a 5-point scale; higher scores indicate greater self-efficacy.
Treatment Expectations and Experiences (Generic Expectation Evaluation Questionnaire) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Treatment-related expectations and experiences assessed with the Generic Expectation Evaluation Questionnaire (G-EEE), including expected symptom improvement, worsening, and side effects prior to treatment, as well as perceived changes during and after treatment.
  Ratings are provided on numerical rating scales from 0 to 10, with higher scores indicating stronger expectations or perceived effects.
Suicidal Ideation and Behavior (Suicide Behaviors Questionnaire-Revised) | Baseline, post-treatment (5 weeks), 3-month and 6-month follow-ups
  Suicidal ideation and behavior assessed with the Suicide Behaviors Questionnaire-Revised (SBQ-R), a 4-item self-report screening instrument covering lifetime suicidal ideation and attempts, frequency of ideation, threat of attempt, and self-assessed likelihood of future suicide.
  Item responses are recoded and summed to yield a total score ranging from 3 to 18; higher scores indicate greater suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (1):
- Philipps-University Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available upon reasonable request after publication of the main results, in accordance with DFG and CRC/TRR 393 data sharing policies. Data access will require a data use agreement and ethical approval.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data and supporting documents will be available within 12 months after publication of the primary outcomes and will remain accessible for at least 10 years thereafter.
Access Criteria: De-identified individual participant data (IPD), study protocol, statistical analysis plan, and informed consent form will be made available to qualified researchers upon reasonable request. Access will be provided via the Open Science Framework (OSF) project page once data are curated and anonymized. Requests for access can be directed to the principal investigators of Project C02 within the CRC/TRR 393. Data will be available for scientific use after publication of the main results.

REFERENCES:
- [Background] Treadway MT, Zald DH. Reconsidering anhedonia in depression: lessons from translational neuroscience. Neurosci Biobehav Rev. 2011 Jan;35(3):537-55. doi: 10.1016/j.neubiorev.2010.06.006. Epub 2010 Jul 11. PMID 20603146
- [Background] Whitton AE, Treadway MT, Pizzagalli DA. Reward processing dysfunction in major depression, bipolar disorder and schizophrenia. Curr Opin Psychiatry. 2015 Jan;28(1):7-12. doi: 10.1097/YCO.0000000000000122. PMID 25415499
- [Background] Watkins E, Brown RG. Rumination and executive function in depression: an experimental study. J Neurol Neurosurg Psychiatry. 2002 Mar;72(3):400-2. doi: 10.1136/jnnp.72.3.400. PMID 11861707
- [Background] Kazdin AE. Mediators and mechanisms of change in psychotherapy research. Annu Rev Clin Psychol. 2007;3:1-27. doi: 10.1146/annurev.clinpsy.3.022806.091432. PMID 17716046
- [Background] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Background] Rief W, Shedden-Mora MC, Laferton JA, Auer C, Petrie KJ, Salzmann S, Schedlowski M, Moosdorf R. Preoperative optimization of patient expectations improves long-term outcome in heart surgery patients: results of the randomized controlled PSY-HEART trial. BMC Med. 2017 Jan 10;15(1):4. doi: 10.1186/s12916-016-0767-3. PMID 28069021
- [Background] Rief W, Anna Glombiewski J. The role of expectations in mental disorders and their treatment. World Psychiatry. 2017 Jun;16(2):210-211. doi: 10.1002/wps.20427. No abstract available. PMID 28498580
- [Background] Potsch L, Rief W. Transdiagnostic considerations of the relationship between reward sensitivity and psychopathological symptoms - a cross-lagged panel analysis. BMC Psychiatry. 2023 Sep 4;23(1):650. doi: 10.1186/s12888-023-05139-3. PMID 37667190
- [Background] Pizzagalli DA. Toward a Better Understanding of the Mechanisms and Pathophysiology of Anhedonia: Are We Ready for Translation? Am J Psychiatry. 2022 Jul;179(7):458-469. doi: 10.1176/appi.ajp.20220423. PMID 35775159
- [Background] Pizzagalli DA. Depression, stress, and anhedonia: toward a synthesis and integrated model. Annu Rev Clin Psychol. 2014;10:393-423. doi: 10.1146/annurev-clinpsy-050212-185606. PMID 24471371
- [Background] Pan PM, Sato JR, Paillere Martinot ML, Martinot JL, Artiges E, Penttila J, Grimmer Y, van Noort BM, Becker A, Banaschewski T, Bokde ALW, Desrivieres S, Flor H, Garavan H, Ittermann B, Nees F, Papadopoulos Orfanos D, Poustka L, Frohner JH, Whelan R, Schumann G, Westwater ML, Grillon C, Cogo-Moreira H, Stringaris A, Ernst M; IMAGEN Consortium. Longitudinal Trajectory of the Link Between Ventral Striatum and Depression in Adolescence. Am J Psychiatry. 2022 Jul;179(7):470-481. doi: 10.1176/appi.ajp.20081180. Epub 2022 May 18. PMID 35582783
- [Background] Kube T, Schwarting R, Rozenkrantz L, Glombiewski JA, Rief W. Distorted Cognitive Processes in Major Depression: A Predictive Processing Perspective. Biol Psychiatry. 2020 Mar 1;87(5):388-398. doi: 10.1016/j.biopsych.2019.07.017. Epub 2019 Jul 29. PMID 31515055
- [Background] Kube T, Rief W, Gollwitzer M, Gartner T, Glombiewski JA. Why dysfunctional expectations in depression persist - Results from two experimental studies investigating cognitive immunization. Psychol Med. 2019 Jul;49(9):1532-1544. doi: 10.1017/S0033291718002106. Epub 2018 Aug 22. PMID 30131084
- [Background] Kirchner L, Rief W, Muller L, Buchwald H, Fuhrmann K, Berg M. Depressive symptoms and the processing of unexpected social feedback: Differences in surprise levels, feedback acceptance, and "immunizing" cognition. PLoS One. 2024 Aug 26;19(8):e0307035. doi: 10.1371/journal.pone.0307035. eCollection 2024. PMID 39186743
- [Background] Insel TR, Cuthbert BN. Medicine. Brain disorders? Precisely. Science. 2015 May 1;348(6234):499-500. doi: 10.1126/science.aab2358. No abstract available. PMID 25931539
- [Background] Hofmann SG, Asnaani A, Vonk IJ, Sawyer AT, Fang A. The Efficacy of Cognitive Behavioral Therapy: A Review of Meta-analyses. Cognit Ther Res. 2012 Oct 1;36(5):427-440. doi: 10.1007/s10608-012-9476-1. Epub 2012 Jul 31. PMID 23459093
- [Background] Greenberg T, Chase HW, Almeida JR, Stiffler R, Zevallos CR, Aslam HA, Deckersbach T, Weyandt S, Cooper C, Toups M, Carmody T, Kurian B, Peltier S, Adams P, McInnis MG, Oquendo MA, McGrath PJ, Fava M, Weissman M, Parsey R, Trivedi MH, Phillips ML. Moderation of the Relationship Between Reward Expectancy and Prediction Error-Related Ventral Striatal Reactivity by Anhedonia in Unmedicated Major Depressive Disorder: Findings From the EMBARC Study. Am J Psychiatry. 2015 Sep 1;172(9):881-91. doi: 10.1176/appi.ajp.2015.14050594. Epub 2015 Jul 17. PMID 26183698
- [Background] Friston K. The free-energy principle: a unified brain theory? Nat Rev Neurosci. 2010 Feb;11(2):127-38. doi: 10.1038/nrn2787. Epub 2010 Jan 13. PMID 20068583
- [Background] Fried EI, Nesse RM. Depression sum-scores don't add up: why analyzing specific depression symptoms is essential. BMC Med. 2015 Apr 6;13:72. doi: 10.1186/s12916-015-0325-4. PMID 25879936
- [Background] Ferrari A, Richter D, de Lange FP. Updating Contextual Sensory Expectations for Adaptive Behavior. J Neurosci. 2022 Nov 23;42(47):8855-8869. doi: 10.1523/JNEUROSCI.1107-22.2022. Epub 2022 Oct 24. PMID 36280262
- [Background] Fazeli S, Buchel C. Pain-Related Expectation and Prediction Error Signals in the Anterior Insula Are Not Related to Aversiveness. J Neurosci. 2018 Jul 18;38(29):6461-6474. doi: 10.1523/JNEUROSCI.0671-18.2018. Epub 2018 Jun 22. PMID 29934355
- [Background] Ewen AI, Bleichhardt G, Rief W, Von Blanckenburg P, Wambach K, Wilhelm M. Expectation focused and frequency enhanced cognitive behavioural therapy for patients with major depression (EFFECT): a study protocol of a randomised active-control trial. BMJ Open. 2023 Mar 22;13(3):e065946. doi: 10.1136/bmjopen-2022-065946. PMID 36948546
- [Background] D'Astolfo L, Rief W. Learning about Expectation Violation from Prediction Error Paradigms - A Meta-Analysis on Brain Processes Following a Prediction Error. Front Psychol. 2017 Jul 28;8:1253. doi: 10.3389/fpsyg.2017.01253. eCollection 2017. PMID 28804467
- [Background] Cuijpers P, Miguel C, Harrer M, Plessen CY, Ciharova M, Ebert D, Karyotaki E. Cognitive behavior therapy vs. control conditions, other psychotherapies, pharmacotherapies and combined treatment for depression: a comprehensive meta-analysis including 409 trials with 52,702 patients. World Psychiatry. 2023 Feb;22(1):105-115. doi: 10.1002/wps.21069. PMID 36640411
- [Background] Cuijpers P, Karyotaki E, Weitz E, Andersson G, Hollon SD, van Straten A. The effects of psychotherapies for major depression in adults on remission, recovery and improvement: a meta-analysis. J Affect Disord. 2014 Apr;159:118-26. doi: 10.1016/j.jad.2014.02.026. Epub 2014 Feb 24. PMID 24679399
- [Background] Beck AT, Haigh EA. Advances in cognitive theory and therapy: the generic cognitive model. Annu Rev Clin Psychol. 2014;10:1-24. doi: 10.1146/annurev-clinpsy-032813-153734. Epub 2014 Jan 2. PMID 24387236
- See also: World Health Organization. (2023). Mental health at work. WHO. — https://www.who.int/news-room/fact-sheets/detail/mental-health-at-work